CLINICAL TRIAL: NCT06521528
Title: A Pilot Clinical Study to Evaluate the Feasibility of Using the Single Patient Classifier as a Prognostic Test in Stage II-III Gastric Cancer Patients.
Brief Title: A Pilot Clinical Study to Evaluate the Feasibility of Using the SPC Test
Status: Active, not recruiting | Type: Observational
Sponsor: Novomics. Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Feasibility Study
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: None Retained — FFPE samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Feasibility cohort: patients who underwent gastrectomy between September 2019 and August 2020 across nine hospitals.
  Interventions: Device: nProfiler I Stomach Cancer Assay Kit

INTERVENTIONS:
Device: nProfiler I Stomach Cancer Assay Kit — nProfiler I Stomach Cancer Assay Kit (Novomics Co., Korea)

SUMMARY:
Precision medicine approaches emphasize the importance of reliable prognostic tools for guiding individualized therapy decisions. In this study, we evaluated the clinical feasibility of the Single Patient Classifier (SPC) test, a new clinical-grade prognostic assay, in stage II-III gastric cancer patients.

DETAILED DESCRIPTION:
A prospective multicenter study was conducted, involving 237 patients who underwent gastrectomy between September 2019 and August 2020 across nine hospitals. The SPC test was employed to stratify patients into risk groups, and its feasibility and performance were evaluated. The primary endpoint was the proportion of the cases in which the test results were timely delivered before selecting postoperative treatment. Furthermore, 3-year disease-free survivals of risk groups were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* being ≥19 years of age
* having a histologically confirmed diagnosis of stage II or III AGC according to the American Joint Committee on Cancer (AJCC) staging system (sixth edition)
* underwent radical gastrectomy without prior neo-adjuvant chemoradiotherapy and did not receive adjuvant chemotherapy
* having no visually or microscopically detectable residual tumors.

Exclusion Criteria:

-Those with insufficient quantity or quality of ribonucleic acid (RNA) for analysis were excluded from the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: histologically confirmed diagnosis of stage II or III AGC
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Timely delivered proportion | 14 days
  the proportion of the cases in which the test results were timely delivered before selecting postoperative treatment

SECONDARY OUTCOMES:
3-year disease free survival of the enrolled patients. | 3-years after the enrollment completion
  Statistical significance (P value of <0.05)
5-year overall survival of the enrolled patients. | 5-years after the enrollment completion
  Statistical significance (P value of <0.05)

CONTACTS AND LOCATIONS:
Overall Officials: Young-Woo Kim, MD., Ph.D, Principal Investigator — National Cancer Center
Locations (1):
- Novomics. Co., Ltd., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided